CLINICAL TRIAL: NCT03499184
Title: Effect of Probiotic Along With Scaling and Root Planing in the Treatment of Chronic Periodontitis
Brief Title: Adjunctive Probiotics in Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin Hospital (Other)
Responsible Party: Principal Investigator, Sana Ikram, MPhil Trainee, Doctor, Lecturer, MPhil trainee, Ziauddin Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0220817SIOB
Record Dates: First submitted 2018-04-03; First posted 2018-04-17 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Chronic Periodontitis; Probiotics
MeSH Terms: conditions — Chronic Periodontitis | interventions — Amoxicillin; Metronidazole; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Local Probiotics (Experimental): P Flor (Lactobacillus reuteri 1.2 billion CFU) will be delivered locally every 12 hours for 12 weeks
  Interventions: Dietary Supplement: P Flor locally delivered
- Systemic Probiotics (Experimental): P Flor (Lactobacillus reuteri 1.2 billion CFU) will be administered every 12 hours for 12 weeks
  Interventions: Dietary Supplement: P Flor systemically administered
- Systemic Antibiotics (Active Comparator): Amoxil 500 mg capsule and Flagyl 400 mg tablet by mouth, will be given every 8 hours for 5 days
  Interventions: Drug: Amoxil 500 mg Oral Capsule; Drug: Flagyl 400 mg Tablet

INTERVENTIONS:
Dietary Supplement: P Flor locally delivered — Locally delivered Lactobacillus reuteri 1.2 CFU per gram
  Arms: Local Probiotics
Dietary Supplement: P Flor systemically administered — Systemically administered Lactobacillus reuteri 1.2 CFU per gram
  Arms: Systemic Probiotics
Drug: Amoxil 500 mg Oral Capsule — Systemically administered Amoxil 500 mg thrice daily
  Arms: Systemic Antibiotics
Drug: Flagyl 400 mg Tablet — Systemically administered Metronidazole 400 mg twice daily
  Arms: Systemic Antibiotics

SUMMARY:
This study will assess clinical and microbiological efficacy of probiotics and antibiotics in patients of chronic periodontitis as an adjunctive to scaling and root planing (SRP) in reducing bacterial count and in improving clinical periodontal parameters over the period of 12 weeks.Also the comparison between these adjunctives will be made for clinical assessment clinical periodontal parameters will be taken .these parameters plaque index (PI), gingival index (GI), clinical attachment loss (CAL) and pocket probing depth (PPD) for microbiological assessment plaque sample will be taken, DNA will be extracted and then sample will be processed through quantitative polymerase chain reaction (qPCR) for quantitative analysis of bacterial count of porphyromonas gingivalis.

DETAILED DESCRIPTION:
In this clinical trial total 60 participants of clinically diagnosed chronic periodontitis will be recruited after taking a written consent for their approval. Participants will be divided into 3 groups A, B and C through the process of randomization using a method of opaque sealed envelopes. A research assistant will be hired for the purpose of randomization and allocation concealment. All participants will be asked to pick an opaque envelope containing the details of treatment products. After randomization plaque sample will be obtained from the depth of periodontal pockets and all the clinical periodontal parameters will be recorded in every participant. Then all the participants will undergo SRP. After SRP group A will be given antibiotics Amoxicillin 500 milligrams (mg) for 3 times a day (TDS) and Metronidazole 400 milligrams (mg) for twice a day (BD) for 5 days. Group B will be given probiotics lactobacillus reuteri 1.2 billion colony forming unit (CFU) sachets twice daily for swallowing with water for 12 weeks. Group C will be given lactobacillus sachets of same amount and participant will be asked to mix it with little amount of water and apply it on teeth with the toothbrush twice daily after brushing with standard tooth paste for 12 weeks. Patients will be recalled at the interval of 3, 6, 9 and 12 weeks for the recording of clinical periodontal parameters. After completion of trial plaque sample will be taken again from every participant and will be processed through qPCR to check bacterial count of porphyromonas gingivalis before and after treatment. Whereas comparison between clinical periodontal parameters will be made at the interval of 0, 3, 6, 9, 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically diagnosed chronic periodontitis with a pocket depth of ≥4mm.
* Patients with age ≥30 years.

Exclusion Criteria:

* Handicapped patients who are physically or mentally unable to maintain their oral hygiene.
* Pregnant and lactating females.
* Patients with habits of smoking, chewing tobacco and alcohol consumption.
* Patients on local or systemic antibiotic treatment.
* Patients with any systemic diseases.
* Patients with the history of any periodontal therapy within last 6 months.
* Patients undergoing orthodontic treatment.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Change in periodontal pocket depth (PPD) | Baseline, 3, 6, 9 and 12 weeks
  It is the distance from tip of free gingival margin to the base of pocket
Change in clinical attachment level (CAL) | Baseline, 3, 6, 9 and 12 weeks
  It is the distance from cementoenamel junction to the base of the pocket around the tooth
Change in bacterial load of Porphyromonas gingivalis | Baseline and 12 weeks after completion of trial
  Bacterial count or the quantity of porphyromonas gingivalis in the sample

SECONDARY OUTCOMES:
Change in the Plaque index (PI) | Baseline, 3, 6, 9 and 12 weeks
  How much surface of tooth is covered by the plaque will be recorded.
Change in Gingival index (GI) | Baseline, 3, 6, 9 and 12 weeks
  Gingival color texture and inflammation will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziauddin Dental College, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided